CLINICAL TRIAL: NCT00612651
Title: A Phase I Trial of the Addition of the Farnesyl Transferase Inhibitor, SCH 66336, to Temodar for Patients With Grade 3 and 4 Malignant Gliomas
Brief Title: PH I Addition of Farnesyl Transferase Inhibitor to Temozolomide for Pts w Gr 3 & 4 Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005027; 7009/Pro00005027 (Other: Duke Institutional Review Board)
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Gliosarcoma; Glioblastoma; Anaplastic Astrocytoma
Keywords: GBM; Malignant glioma; Brain tumor; Temodar; Temozolomide; SCH 66336; Farnesyl transferase inhibitor; Glioblastoma multiforme; Gliosarcoma; Anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligoastrocytoma
MeSH Terms: conditions — Gliosarcoma; Glioblastoma; Astrocytoma; Glioma; Brain Neoplasms; Oligodendroglioma | interventions — Temozolomide; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enzyme-inducing anti-epileptic drugs (EIAEDs) (Other): Patients receiving enzyme-inducing anti-epileptic drugs (EIAEDs)such as carbamazepine, phenobarbitol, phenytoin, phosphenytoin, oxcarbamazepine, primadone)
  Interventions: Drug: Temodar and SCH 66336
- no enyzme-inducing anti-epileptic drugs (Other): Patients on non CYP3A4-inducing anti-convulsants or patients not on any anti-convulsants.
  Interventions: Drug: Temodar and SCH 66336

INTERVENTIONS:
Drug: Temodar and SCH 66336 — 2 separate strata accrued independently: Stratum 1-pts receiving CYP3A4-inducing anticonvulsants. Stratum 2-pts on non CYP3A4-inducing anticonvulsants or pts not on any anti-convulsants. Each strata treated & escalated independent of each other. Temozolomide administered orally at dose of 150 mg/m2 daily for 5 days, at bedtime, for 1st cycle & escalated to 200 mg/m2 daily for 5 days, at bedtime during subsequent cycles if tolerated. Treatment cycles repeated every 4wks following doses of Temozolomide from previous cycle. SCH 66336 administered orally twice daily, approximately every 12hrs. Except as specifically noted, pts advised to take capsules wh morning & evening meals, with approximately 240ml of non-carbonated water. Initial doses will be 125mg BID for stratum 1 & 75mg BID for stratum2. Treatment cycles repeated every 4 wks following dose of Temozolomide from previous cycle.
  Other Names: Temodar-Temozolomide; Farnesyl transferase inhibitor-SCH 66336

SUMMARY:
Objectives:

To determine maximum tolerated dose of farnesyl transferase inhibitor, SCH 66336, when administered w TEMODAR®.

To characterize any toxicity associated w combo of farnesyl transferase inhibitor, SCH 66336, & TEMODAR®.

To observe patients for clinical antitumor response when treated with combination of farnesyl transferase inhibitor, SCH 66336, & TEMODAR®.

To assess pharmacokinetics of SCH 66336 for patients on & not on enzyme inducing antiepileptic drugs.

DETAILED DESCRIPTION:
2 separate strata accrued independently of each other: Stratum1-Patients receiving Dilantin, Tegretol / phenobarbital. Stratum2-Patients on anti-convulsants other than Dilantin, Tegretol / phenobarbital / Patients not on any anti-convulsants. Each stratum treated & escalated independent of each other. Temozolomide administered orally at dose of 150mg/m2 daily for 5 days, at bedtime, for 1st cycle & escalated to 200mg/m2 daily for 5 days, at bedtime during subsequent cycles if tolerated. Treatment cycles may be repeated every 4 weeks following doses of Temozolomide from previous cycle. SCH 66336 administered orally twice day, approximately every 12hrs. Initial doses will be 125mg BID for stratum 1 & 75mg for stratum 2. Treatment cycles may be repeated every 4 weeks following dose of Temozolomide from previous cycle.

Subjects are patients with malignant glioma histologically confirmed at diagnosis, who were treated previously with conventional external beam radiation (XRT) & with or without chemo, & have stable disease, recurrence/relapse at time of enrollment. Approximately 48 subjects will be enrolled.

Temozolomide has been well tolerated by both adults & children with most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea & vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, & hepatotoxicity. Hypersensitivity reactions have not yet been noted with Temozolomide. As is case with many anti-cancer drugs, Temozolomide may be carcinogenic. Rats given Temozolomide have developed breast cancer. Significance of this finding for humans is not presently known.

Significant adverse events observed for SCH66336 have included vomiting, diarrhea, anorexia, headaches, reversible renal toxicities, & hematological toxicities. SCH 66336, although not genotoxic, inhibits rapidly proliferating cells & at high doses inhibits spermatogenesis in male rats. It is not clear that inhibition of spermatogenesis is reversible,& patients should be advised of possibility of irreversible sterility.

ELIGIBILITY:
Inclusion Criteria:

* Pts with MG histologically confirmed at diagnosis, who were treated previously with conventional external beam radiation & with or without chemotherapy, & have stable disease, recurrence or relapse at the time of enrollment.
* Age > or = to 18 years.
* Patients who have had previous surgical resection(s) are eligible.
* Interval of at least 3 weeks between prior surgical resection, 2 weeks between prior radiotherapy, or 4 weeks between prior chemotherapy, unless there is unequivocal evidence of tumor progression after surgery, radiotherapy, or chemotherapy.
* Karnofsky performance score > or = to 60%.
* Adequate hematologic, renal & liver function as demonstrated by lab values performed within 14 days, inclusive, prior to administration of chemotherapy:
* ANC > or = to 1500/mm3
* Platelet count > or = to 100,000/mm3
* Hemoglobin > or = to 10 gm/dL
* BUN and serum creatinine <1.5 times upper limit of lab normal
* Total serum bilirubin <1.5 times upper limit of lab normal
* SGOT <2.5 times upper limit of lab normal
* Patients must have recovered from any effects of major surgery.
* Patients must have life expectancy of greater than 12 weeks.
* Patients or legal guardian must give written, informed consent.

Exclusion Criteria:

* Patients requiring immediate radiation therapy.
* Patients who have not recovered from surgery.
* Patients who are not neurologically stable for 2 weeks prior to study entry.
* Patients who are poor medical risks because of non-malignant systemic disease as well as those with acute infection treated with intravenous antibiotics.
* Frequent vomiting or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction).
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Known HIV positivity or AIDS-related illness.
* Pregnant or nursing women.
* Women of childbearing potential who are not using an effective method of contraception. Women of childbearing potential must have a negative serum pregnancy test 72 hours prior to administration of study drug and be practicing medically approved contraceptive precautions.
* Men who are not advised to use an effective method of contraception.
* Patients taking immuno-suppressive agents other than prescribed corticosteroids.
* Patients previously treated with farnesyl transferase inhibitors.
* Patients with significant QTc prolongation (>500 msec)as evaluated by an EKG.
* Patients having presented prior disease progression on TEMODAR.
* Patients having presented any grade 4 hematologic toxicity or grade 3 or 4 non-hematologic toxicity on TEMODAR in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/